CLINICAL TRIAL: NCT05033899
Title: Enhanced Recovery After Spinal Surgery Protocol Versus Conventional Care in Non Insulin Diabetic Patients:A Prospective Randomized Study
Brief Title: Enhanced Recovery After Spinal Surgery Protocol Versus Conventional Care in Non Insulin Diabetic Patients ( ERAS )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, sarah mohamed, Assistant lecturer, alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ERAS diabetic spine surgery
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: ERAS; Surgery; Non Insulin Dependent Diabetes Mellitus; Lumbar Spine Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Spinal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group E: ERAS group (Experimental): 36 non-insulin dependent diabetic patients will undergo lumbar decompression surgery following ERAS protocol.
  Interventions: Other: ERAS protocol
- group C: conventional group (No Intervention): conventional perioperative care.

INTERVENTIONS:
Other: ERAS protocol — to compare between Enhanced Recovery After Surgery (ERAS) protocol and conventional care in non-insulin dependent diabetic patients undergoing lumbar spine surgery.
  Other Names: enhanced recovery after surgery protocol
  Arms: group E: ERAS group

SUMMARY:
enhanced recovery after spinal surgery protocol (ERAS) versus conventional care in non insulin diabetic patients. Our hypothesis is that non-insulin dependent diabetic patients who will undergo lumbar decompression surgery following ERAS care may have higher quality of recovery after surgery, lower postoperative pain scores, decreased opioid consumption, reduced Length of stay and reduce perioperative stress compared to conventional general anaesthesia.

DETAILED DESCRIPTION:
72 patients of American Society of Anaesthesiology (ASA) physical status II or III, of both sexes, aged (30-65) years admitted to department of neurosurgery, Alexandria Main University Hospital and scheduled for elective lumbar decompression surgeries under the effect of general anaesthesia.

All patients will be randomized 1:1 using a sealed envelope method to receive their perioperative care under our ERAS protocol versus conventional care. The envelope will be opened by an observer not involved in the study. Patients will be divided into two equal groups.

Group (E): ERAS group: 36 non-insulin dependent diabetic patients will undergo lumbar decompression surgery following ERAS protocol.

Group (C): Conventional group: 36 non-insulin dependent diabetic patients will undergo lumbar decompression surgery under conventional perioperative care.

During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes, fasting blood glucose, glycosylated haemoglobin (HBA1C), liver function tests and any other investigation needed.

Pre-anaesthetic preparation and premedication:

In both groups:

Every patient will be informed about the ERAS protocol and the procedure of US guided erector spinae plane block.

Informed written consent, from all individual participants who will be included in this study or their legal representatives will be taken during preoperative visit.

The patient should be trained during preoperative visit on a visual analogue scale (VAS), with 0 corresponding to no pain and 10 to the worst pain imaginable.

Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery.

Oral hypoglycemic control drugs will be discontinued after the last meal. In ERAS group, patients will receive solid foods until 6 hours before surgery and clear fluids until 4 hours prior. A 400 ml of clear carbohydrate-rich beverage (12.5g/100ml) will be supplied before the day of surgery, to be consumed 4 hours before the scheduled time of surgery, while in non- ERAS group, patients will fast for 8 hours.(25) In both groups, Antibiotic prophylaxis (ceftriaxone 2 g intravenously) will be given 1 hour before surgical incision.

In ERAS group, Oral pre-emptive analgesia will be provided in the holding area on the day of surgery, and will include acetaminophen (1000 mg), gabapentin (300 mg), provided there is no contraindications, while in non- ERAS group, no analgesia will be given.

Finger stick glucose monitoring will be applied every 2 hours and rapid acting subcutaneous insulin will be given if blood glucose is > 180 mg/dl.

On arrival to operative theatre, before the induction of anaesthesia, standard monitoring will be established using multichannel monitor (Carescape Monitor B650, General electric (GE) Healthcare Finland) to monitor the following in both groups:

Electrocardiogram (ECG) for heart rate and rhythm. (Beats/min). Non-invasive measurement of arterial blood pressure. (Mean blood pressure in mmHg).

Pulse oxygen saturation. (SpO2%). End tidal carbon dioxide ( CO2) tension (in mmHg). Entropy Neuromuscular transmission (TOF; transmission with four stimuli) Nasopharyngeal core temperature In ERAS group, the non-invasive cardiac output monitoring device (ICON, Osypka Medical, Berlin, Germany) will be attached to the patient by four electrodes. Two electrodes will be on the right side of the neck, the two other electrodes on the left side of the chest opposite to the xiphoid process at the mid axillary line.

Anaesthesia:

After preoxygenation for 3 minutes, anaesthesia will be induced in both groups with propofol 0.5-2mg/kg until loss of verbal response, fentanyl 2µg/kg and atracurium 0.5 mg/kg intravenously. Anaesthesia will be maintained by isoflurane with 50% oxygen in air (1.2-1.5 %) to maintain entropy between 40-60. Mechanical ventilation will be performed with a constant tidal volume of 8 ml/ kg and a respiratory rate of 10 to 12 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 per cent with 50 percent oxygen in air. Incremental doses of atracurium will be given according to nerve stimulator.

In both groups, signs of insufficient analgesia (eg, tachycardia over 20% of the preoperative value occur during anaesthesia) or somatic response (eg, movement ,tearing ,or sweating), will be treated with additional boluses of fentanyl 0.5 mcg/kg intraoperatively as needed. Strategies to prevent hypothermia include the use of warmed infusion liquids, and forced air-warming blankets will be done to avoid intraoperative hypothermia.

In ERAS group, dual antiemetic prophylactic therapy (metoclopramide 10 mg iv. and dexamethasone 8mg iv) will be administered intravenously immediately after induction. Also, intravenous infusion of tranexamic acid 10 mg/kg(27) will be given in this group.

In ERAS group, after turning the patient into prone position, US guided erector spinae plane (ESP) block will be given.

In both groups: Intraoperative blood glucose level will be maintained intraoperatively between 140 and 180 mg/dl. If a patient has a blood glucose level greater than or equal to 180, an IV insulin drip will be initiated. Starting dose of insulin drip (units/hour) can be calculated with blood glucose/100 and titrated according to the following regimen by checking the blood glucose level every hour.

At the end of the surgery, patient will be turned to supine position then anaesthesia will be discontinued and 100% oxygen will be administered then the oral secretions will be aspirated. The residual neuromuscular relaxation will be reversed using neostigmine 40 ug/kg and atropine 20 ug/kg slowly by the intravenous route. Extubation will be performed awake after the return of protective airway reflexes.

Upon admission to the post-anesthesia care unit (PACU), all patients will be observed continuously for at least 30 min by observers blinded to study groups.

All the procedures will be performed by the same three surgeons, all with a clinical experience of more than 5 years using the same surgical technique for each type of surgery. Due to the requirement for active patient participation, it will not possible to perform the study with blinded participants and care providers. Only those who will collect and assess the postoperative outcomes in PACU and the ward will be blinded to the patient group assignment and to the nature of the study.

Postoperative Management:

In ERAS group, immediate postoperative management will include cessation of intravenous fluid administration, oral intake, and mobilization within 2 hours of PACU arrival.

In ERAS group, target postoperative glycemic range will be between 140 and 180mg/dl. The insulin infusion will be continued postoperatively until oral intake will be established, after which the preoperative diabetes treatment will be resumed. The first dose of the oral hypoglycemic drugs will be given 30-60 min before disconnecting the infusion.

In both groups, intravenous paracetamol 1 g/6 hours (Perfalgan® 100 ml vial The Union of applied scientific pharmacology (UPSA) France) and intravenous ketorolac loading 30 mg then 15mg/8 hours regularly will be given for postoperative pain relief. Nalbuphine 0.15 mg/kg IV will be given as postoperative rescue analgesia if VAS was ≥ 4. The incidence of postoperative nausea and vomiting (PONV) will be assessed by a nurse for the first 24 hrs and only 2 possible answers will be accepted (yes or no).

The volume status will be assessed by the blood pressure, heart rate, urine output and mental status of patients. Patients will be discharged from the PACU according to modified Aldrete score (if the score is ≥ 9, the patient can be discharged).

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-65 years, both sexes
* ASA physical status class II and III
* 2-3 levels elective lumbar surgery.
* Controlled non- insulin dependent diabetic patients (HbA1C ≤ 7% )

Exclusion Criteria:

* Cervical and thoracic surgery
* More than 3 levels surgery.
* Cognitive impairment.
* Infection, trauma, neoplasm.
* Revision surgery.
* Patients with BMI > 35 kg/m2, renal or cardiac and liver failure.
* Patients with retinopathy or reduction of visual acuity.
* Patients with known hypersensitivity or contraindication to medications.
* Coagulopathy or uncontrolled Diabetes mellitus (DM) .
* Patients receiving any analgesic medications within 24 h pre-operative or antiplatelet medication within the past 1 week.
* Patients who had symptoms of nausea and vomiting or received an antiemetic within 24 h of surgery.
* Random blood glucose more than 250 mg/dl just before shifting the patient from the ward to the operating room.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of recovery after surgery (QoR40) | postoperative day 2
  40-item questionnaire that assesses five dimensions of recovery after surgery and anesthesia: comfort, emotions, physical independence, patient support, and pain and has a mean time to completion of 5 min.

SECONDARY OUTCOMES:
heart rate | surgery period
  beats/minute
mean arterial blood pressure | surgery period
  mmHg
Postoperative pain score | 8 hours postoperative
  Scale of 0-10, 0 being no pain, 10 being the worst pain possible
Perioperative nalbuphine requirements | 24 hours postoperative
  measured in mg
postoperative hospital stay | postoperative day 5
  measured in days after surgery
Time to first postoperative analgesic request | 24 hours postoperative
  measured in minutes
Blood sugar level | time of admission to PACU
  mg/dl
Number of patients required rescue anti-emetic postoperatively | 24 hours postoperative
  patients receive ondansetron
number of participants with Perioperative complications | postoperative day 5
  vomiting, wound infection, urinary tract infection , deep vein thrombosis, haematoma
serum markers of stress response: C reactive protein ( CRP) | postoperative day 2
  mg/dl
serum markers of stress response: interleukin 6 ( IL-6) | postoperative day 2
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: ashraf arafat, MD, Study Director — Alexandria University; Emad Abdelmoneim arida, MD, Study Director — Alrxandria university; Rania Aboelfetouh, MD, Study Director — Alexandria University; Abdulrahman Elhabashy, MD, Study Director — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
through clinical trials
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months up to 1 year
Access Criteria: ERAS, lumbar spine surgery, non insulin diabetic patients, quality of recovery

REFERENCES:
- [Background] Soffin EM, Beckman JD, Tseng A, Zhong H, Huang RC, Urban M, Guheen CR, Kim HJ, Cammisa FP, Nejim JA, Schwab FJ, Armendi IF, Memtsoudis SG. Enhanced Recovery after Lumbar Spine Fusion: A Randomized Controlled Trial to Assess the Quality of Patient Recovery. Anesthesiology. 2020 Aug;133(2):350-363. doi: 10.1097/ALN.0000000000003346. PMID 32433277